CLINICAL TRIAL: NCT00621179
Title: Do Endometrial Implantation Markers Predict in Vitro Fertilization-embryo Transfer Cycle Outcomes in Endometriosis Patients Pretreated With Leuprolide Acetate in Depot Suspension?
Brief Title: Endometrial Markers and Response of Endometriosis Patients to Prolonged GnRH Agonist Prior to IVF
Acronym: IntegrinIVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colorado Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Eric Surrey, M.D., Medical Director, Colorado Center for Reproductive Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IntegrinIVF
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis; Infertility
Keywords: Endometriosis,infertility,in vitro fertilization
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Positive endometrial alpha v, beta 3 vitronectin expression. Standard controlled ovarian stimulation protocol followed by in vitro fertilization Intervention: No intervention
  Interventions: Other: No intervention
- Group 2 (Experimental): Intervention: Positive endometrial alpha v beta 3 vitronectin expression, 3 months of leuprolide acetate in depot suspension administration prior to initiation of controlled ovarian stimulation followed by in vitro fertilization
  Interventions: Drug: Leuprolide acetate in depot suspension
- Group 3 (Experimental): Negative endometrial alpha v, beta 3 vitronectin and administration of leuprolide acetate in depot suspension for 3 months prior to initiation of controlled ovarian stimulation
  Interventions: Drug: Leuprolide acetate in depot suspension
- Group 4 (Active Comparator): Negative endometrial alpha v, beta 3 vitronectin expression and standard controlled ovarian stimulation protocol followed by in vitro fertilization. Intervention: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Leuprolide acetate in depot suspension — Leuprolide acetate in depot suspension 3.75 mg intramuscularly every 28 days x 3
  Other Names: Depot Lupron
  Arms: Group 2; Group 3
Other: No intervention
  Arms: Group 1; Group 4

SUMMARY:
This prospective randomized trial evaluates whether one can predict which infertile women with endometriosis who are candidates for in vitro fertilization will benefit from prolonged therapy with a GnRH agonist by the determination of the absence of endometrial expression of the integrin, alpha v, beta 3 vitronectin. This is a prospective randomized trial in which all patients will undergo endometrial biopsy prior to initiation of ovarian stimulation for in vitro fertilization and then undergo randomization to a three month course of a depot preparation of the GnRH agonist leuprolide acetate in depot suspension prior to ovarian stimulation or standard therapy. prio

DETAILED DESCRIPTION:
See summary

ELIGIBILITY:
Inclusion Criteria:

* Infertility
* Surgical diagnosis of endometriosis
* Normal ovarian reserve testing
* Regular menses

Exclusion Criteria:

* Irregular menses
* Undiagnosed abnormal uterine bleeding
* Pregnancy
* Prior adverse reaction to any GnRH agonist
* Ovarian cystic or solid mass > 3cm in mean diameter at study entry
* Use of a depot preparation of a GnRh agonist or any hormonal therapy for endometriosis within 6 months of study entry
* Current hepatic, renal, hematologic or psychiatric disorder

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2003-03; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Surrey, M.D., Principal Investigator — Colorado Center for Reproductive Medicine
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

REFERENCES:
- [Background] Surrey ES, Silverberg KM, Surrey MW, Schoolcraft WB. Effect of prolonged gonadotropin-releasing hormone agonist therapy on the outcome of in vitro fertilization-embryo transfer in patients with endometriosis. Fertil Steril. 2002 Oct;78(4):699-704. doi: 10.1016/s0015-0282(02)03373-3. PMID 12372443
- [Background] Lessey BA, Castelbaum AJ, Sawin SW, Buck CA, Schinnar R, Bilker W, Strom BL. Aberrant integrin expression in the endometrium of women with endometriosis. J Clin Endocrinol Metab. 1994 Aug;79(2):643-9. doi: 10.1210/jcem.79.2.7519194.
- [Derived] Surrey ES, Lietz AK, Gustofson RL, Minjarez DA, Schoolcraft WB. Does endometrial integrin expression in endometriosis patients predict enhanced in vitro fertilization cycle outcomes after prolonged GnRH agonist therapy? Fertil Steril. 2010 Feb;93(2):646-51. doi: 10.1016/j.fertnstert.2008.12.023. Epub 2009 Jan 26. PMID 19171333

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Positive endometrial alpha v, beta 3 vitronectin expression. Standard controlled ovarian stimulation protocol
- Group 2: Intervention: Positive endometrial alpha v beta 3 vitronectin expression, 3 months of leuprolide acetate in depot suspension administration prior to initiation of controlled ovarian stimulation
- Group 4: Negative endometrial alpha v, beta 3 vitronectin expression and standard controlled ovarian stimulation protocol.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 12 | 8 | 7 | 10
Completed | 12 | 8 | 6 | 9
Not Completed | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Positive endometrial alpha v, beta 3 vitronectin expression. Standard controlled ovarian stimulation protocol followed by in vitro fertilization
- Group 4: Negative endometrial alpha v, beta 3 vitronectin expression and standard controlled ovarian stimulation protocol followed by in vitro fertilization.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 12 | 8 | 7 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 7 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (4.11) | 33.0 (3.55) | 33.86 (2.79) | 32.67 (4.95) | 33.33 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 7 | 9 | 36
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 7 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Responded to Controlled Ovarian Hyperstimulation
Description: Number of patients who responded to controlled ovarian stimulation as evidenced by implantation of embryo. Implantation confirmed by ultrasound at 6 1/2 weeks of pregnancy.
Time Frame: Evaluated at 6 1/2 weeks of pregnancy which is 4 weeks post embryo transfer.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Positive endometrial alpha v, beta 3 vitronectin expression. Standard controlled ovarian stimulation protocol followed by in vitro fertilization Intervention: No intervention
  No intervention
- Group 4: Negative endometrial alpha v, beta 3 vitronectin expression and standard controlled ovarian stimulation protocol followed by in vitro fertilization. Intervention: No intervention
  No intervention
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 12 | 8 | 6 | 9
Participants | 7 | 5 | 3 | 5

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No